CLINICAL TRIAL: NCT04362098
Title: The Effects Over Early Brain Development of a Nurse Home Visitation Program for Pregnant Youth and Their Families Living in a Poor Urban Area in São Paulo, Brazil II
Brief Title: A Home Visiting Program for Pregnant Youth to Promote Early Brain Development II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016/22455-8
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Child Development
Keywords: Child Development; Infant; Mother-Child Relations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse home visits (Experimental): Nurse home visits biweekly.
  Interventions: Behavioral: Home visiting Program for Young Pregnant Women
- Usual care (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Home visiting Program for Young Pregnant Women — The visitation program was elaborated based in the following theoretical principles: a) Albert Bandura's self-efficacy theory; b) Urie Brofenbrenner's bioecological theory, which recognizes the importance of the insertion of individuals in families in varied contexts of life in society; c) John Bowlby and Mary Ainsworth's attachment theory. The basic premises of the intervention are health care, environmental health, life course development, development of parenting ability, relationship with friends and family, and social service support.
  Arms: Nurse home visits

SUMMARY:
Home visiting programs for pregnant women aiming to improve mother-infant relationship has received worldwide attention in the past 30 years. These programs are considered an important strategy to improve women's health during pregnancy, aside from improving child's birthing conditions and allowing parents access to tools which will nurture and properly stimulate their baby, thus promoting emotional and cognitive development. Objectives: The "Nurse home visitation program for pregnant youth" aims to promote infant´s healthy development, from pregnancy to the first months of life, in a high-risk population. Methods: Eighty young pregnant women aged between 14 and 21 years were randomly allocated to the intervention or to usual prenatal care program. The "Nurse home visitation program for pregnant youth" was developed based on Albert Bandura's theory of self-efficacy, on Urie Bronfenbrenner´s bioecological model, which recognizes the importance of individual and family inclusion in various contexts of social life, on John Bowlby and Mary Ainsworth evolutionary theories of attachment, which involves the care practitioner addressing issues such as environmental health, life course and parenting, bond between mother and infant, and infant´s social and cognitive development. Neuropsychomotor development will be assessed at 3, 6, 12 and 24 months using the Bayley Scale of Infant Development. Brain development will be assessed via electroencephalography at 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Low socioeconomic status
* Mother's age between 14-19
* Mother being a primapara
* Gestation between the 8th and 16th week

Exclusion Criteria:

* High-risk gestation
* Mother's Intellectual, visual or auditory disability

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychomotor Development During First Year of Life: Cognition | From 3 to 12 months of age
  Complete child assessment with the Bayley Scale of Infant Development at 3, 6 and 12 months of age.
Change in Neuropsychomotor Development During First Year of Life: Receptive Language | From 3 to 12 months of age
  Child assessment with the Bayley Scale of Infant Development.
Change in Neuropsychomotor Development During First Year of Life: Expressive Language | From 3 to 12 months of age
  Child assessment with the Bayley Scale of Infant Development
Change in Neuropsychomotor Development During First Year of Life: Fine Motor | From 3 to 12 months of age
  Child assessment with the Bayley Scale of Infant Development, fine motor scale.
Change in Neuropsychomotor Development During First Year of Life: Gross Motor | From 3 to 12 months of age
  Child assessment with the Bayley Scale of Infant Development

SECONDARY OUTCOMES:
Change in Child Brain Maturation | At 6 and 12 months
  Assessment of brain wave patterns (alpha, gamma and theta frequencies) via electroencephalography (EEG).
Mother-child Attachment Biomarker | At 6 and 12 months
  Assessment of event-related potential associated with child face recognition of the mother via electroencephalography (EEG).

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme V Polanczyk, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil